CLINICAL TRIAL: NCT04812990
Title: A Cross Sectional Observational Study on Relation Between Oral Manifestation and Hepatitis C in Egypt
Status: Completed | Type: Observational
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Radwa Elsherif, LECTURER, Misr University for Science and Technology
Other Study IDs: HC IN EGYPT
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hepatitis C; Oral Manifestations; in Egyptian Population
MeSH Terms: conditions — Hepatitis C; Oral Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- hepatitis c patients: 50 patients will be recruited for study group from consecutive patients previously diagnosed by hepatitis C regardless of the etiology of the condition and regularly attending at Soad Kafay hospital. Participants with history of smoking and alcoholism that could affect their oral health status were excluded.
- clinically healthy patients: populations will be randomly recruited from the out-patient of dental diagnosis clinic in Misr University For science & technology university to include total 50 clinically healthy participants, with no history of liver disease, or any other chronic debilitating illness, or habit of smoking or drinking, , as well as history of an intervention or condition that could affect the oral mucosa (e.g., history of radiotherapy and/or not receiving any medication that could affect oral health.

SUMMARY:
Hepatitis C virus (HCV) is the major cause of chronic liver disease and has a long-term resultant complications4 and it considered as a major endemic medical health problem in Egypt. It affects multiple organs and reflect various manifestations on oral cavity.The purpose of this study is to assess the prevalence of oral mucosa conditions, type of oral manifestation and gingival lesions in patients with hepatitis C

DETAILED DESCRIPTION:
Study design: It is a cross sectional observational study. Sample size estimation: 100 patients (50 in each groups) A total of 100 adult participants of both genders above 18 years will be included in the study, patients was able and willing to participate in the study. 50 patients will be recruited for study group from consecutive patients previously diagnosed by hepatitis C regardless of the etiology of the condition and regularly attending at Soad Kafay hospital. Participants with history of smoking and alcoholism that could affect their oral health status were excluded. The control group populations will be randomly recruited from the out-patient of dental diagnosis clinic in Misr University For science & technology university to include total 50 clinically healthy participants, with no history of liver disease, or any other chronic debilitating illness, or habit of smoking or drinking, , as well as history of an intervention or condition that could affect the oral mucosa (e.g., history of radiotherapy and/or not receiving any medication that could affect oral health.

Changes in the oral cavity was recorded on the entire mucosal surface recording signs, symptoms, and oral lesion absence or presence. All the information will be recorded and the data will be analyzed after the end of the study . The prevalence of various oral manifestations in hepatitis C patients will be documented.

ELIGIBILITY:
Inclusion Criteria:

* patients previously diagnosed with hepatits c, with education, ability and willing to participate in the study

Exclusion Criteria:

* Patients with systemic diseases such as nutritional deficiency; cardiovascular, respiratory, metabolic, and endocrinal disorders; also smoking and alcoholism that could affect their oral health status were excluded. As well as history of an intervention or condition that could affect the oral mucosa (e.g., history of radiotherapy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hepatic (virus C) and non hepatic patients on Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
oral lesion relation to hepatitis c | six months
  the prevalence to oral lesions related to hepatitis C patients

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry at MUST, Giza, Egypt